CLINICAL TRIAL: NCT01446081
Title: A Phase II Exercise RCT for AML Patients Undergoing Induction Chemotherapy
Brief Title: An Exercise Trial for Acute Myeloid Leukaemia (AML) Patients Undergoing Induction Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AML 003
Record Dates: First submitted 2011-08-04; First posted 2011-10-04 (Estimated); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Acute Myeloid Leukemia
Keywords: chemotherapy; exercise; quality of life; cancer-related fatigue; elderly; physical fitness
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise (Experimental): Patients will receive an individualized, supervised mixed-modality exercise program created by a CSEP-Certified Exercise Physiologist (CEP).
  Interventions: Behavioral: Exercise
- Control (No Intervention): Participants assigned to this arm will receive usual care.

INTERVENTIONS:
Behavioral: Exercise — Patients will receive an individualized, supervised mixed-modality exercise program created by a CSEP-Certified Exercise Physiologist (CEP). They will perform 30 minutes of light to moderate intensity exercise 4-5 times/week tailored to ability. Aerobic exercise will primarily consist of walking and/or stationary cycling. Resistance exercises will target large muscle groups using dumbbells, resistance bands, and stability balls. The CEP will monitor and document details of each exercise session as well as patient tolerance and symptoms, and make appropriate adaptations to ensure program safety and progression. Exercise intensity and duration will vary based on patient tolerance, symptoms and blood parameters. Exercise equipment will be carefully sanitized between each use.
  Arms: Exercise

SUMMARY:
Reduced quality of life, fatigue, and loss of physical function are common in patients getting chemotherapy for acute myeloid leukaemia (AML). The investigators completed a pilot study showing that exercise during active chemotherapy for AML is feasible, safe, and may improve symptoms and physical function. The investigators now propose to compare our hospital-based supervised exercise program to usual care to see if exercise can improve symptoms, physical function, and improve treatment tolerability.

DETAILED DESCRIPTION:
Acute myeloid leukaemia (AML) is a life-threatening malignant blood disorder. Curative treatment requires multiple cycles of intensive chemotherapy. The first cycle, induction, is the most intense and intended to achieve complete disease remission (CR). Induction therapy requires 4-6 weeks of inpatient admission and is associated with extended bed rest and multiple toxicities, leading to physical deconditioning. Regular exercise during induction may reduce declines in physical fitness, leading to improved quality of life (QOL), reduced fatigue, improved tolerance of chemotherapy, and potentially greater survival. Four prior studies of exercise in AML patients undergoing induction have suggested improvements in QOL, fatigue, physical function, and treatment tolerability. However, all 4 studies suffered from major limitations including small sample sizes, design limitations, generalizability concerns, and limited safety information. The investigators conducted a pilot non-randomized study in 35 AML patients and demonstrated feasibility, safety, and potential improvements in QOL, fatigue, and physical fitness outcomes. The investigators now propose a rigorous evaluation of the intervention in a phase II randomized controlled trial (RCT).

Primary objectives include: (1) To determine the efficacy of a supervised mixed-modality exercise program during induction chemotherapy on QOL and fatigue; (2) To determine the efficacy on physical fitness. Our secondary objective is to determine the efficacy on AML treatment tolerability (hospital length of stay, development of sepsis, intensive care unit (ICU) admission, delays in consolidation chemotherapy).

ELIGIBILITY:
Inclusion Criteria:

* Is ≥ 18 years old
* Has newly diagnosed AML, or relapsed AML after having been in CR for at least 6 months
* Is initiating induction chemotherapy
* Is ambulatory without need for human assistance
* Has consented to study
* Is medically cleared for participation by the attending physician

Exclusion Criteria:

* Has another active malignancy
* Has life expectancy < 1 month, physician determined
* Has significant comorbidity
* Has uncontrolled pain
* Has haemodynamic instability
* Lacks fluency in reading and writing English, and there is no translator available for each visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2011-06; Primary Completion 2013-04 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline in quality of life at weeks 4-6 (post-induction) and weeks 10-12 (post-consolidation 1) (QOL) | Baseline (within 5 days of starting chemo), Post-induction (weeks 4-6), Post-consolidation (weeks 10-12)
  EORTC QLQ-C30 (questionnaire)
Change from baseline in fatigue at weeks 4-6 (post-induction) and weeks 10-12 (post-consolidation 1) | Baseline (within 5 days of starting chemo), Post-induction (weeks 4-6), Post-consolidation (weeks 10-12)
  FACT-F (questionnaire)
Change from baseline in fitness measures at weeks 4-6 (post-induction) and weeks 10-12 (post-consolidation 1) | Baseline (within 5 days of starting chemo), Post-induction (weeks 4-6), Post-consolidation (weeks 10-12)
  The fitness assessment will encompass various measures to assess physical fitness. The following measures will be completed: VO2 peak (a measure of aerobic capacity), 6-minute walk test, grip strength and maximal leg strength, chair stands.

SECONDARY OUTCOMES:
Treatment tolerability | Post-induction (weeks 4-6), Post-consolidation (weeks 10-12)
  Length of stay (as an in-patient), development of sepsis (during induction chemotherapy), ICU admission (during induction chemotherapy), delay in consolidation chemotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Shabbir Alibhai, MD, MSc, Principal Investigator — University Health Network, Toronto
Locations (1):
- Princess Margaret Hospital, Toronto, Ontario, Canada